CLINICAL TRIAL: NCT01007292
Title: A Phase II, Multicenter, Open-Label Study Of YM155 Plus Rituximab In Previously Treated Subjects With CD20-Positive B Cell Non-Hodgkin's Lymphoma Who Are Ineligible For Or Have Previously Received An Autologous Stem Cell Transplant
Brief Title: A Study of YM155 Plus Rituximab in Subjects With Non-Hodgkin's Lymphoma Who Have Received Prior Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-031
Record Dates: First submitted 2009-09-24; First posted 2009-11-04 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; relapsed; CD20-Positive; YM155
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — sepantronium; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YM155 plus rituximab (Experimental)
  Interventions: Drug: YM155; Biological: Rituximab

INTERVENTIONS:
Drug: YM155 — intravenous infusion
Biological: Rituximab — intravenous infusion
  Other Names: Rituxan; Mabthera

SUMMARY:
The purpose of this study is to evaluate response rate, survival, safety and tolerability of YM155 given in combination with rituximab in subjects with Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
This is an outpatient study. All subjects enrolled in this study will receive YM155 and rituximab given during 14 day cycles. Each subject will be assessed at the end of each cycle to determine if he or she may continue to the next cycle. Each subject will be eligible to continue receiving the combination regimen in this study until one of the discontinuation criteria is met.

If a subject discontinues treatment without progressive disease (PD) that subject will complete follow-up visits every 12 weeks for 1 year or until initiating another systemic anti-lymphoma treatment, exhibiting PD, or death.

Each subject will be contacted by the study site every 12 weeks for survival following the End of Treatment Visit. The contacts will continue until death or for no more than 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Any stage, histologically confirmed CD20-positive primary or transformed diffuse large B cell lymphoma (DLBCL)or grade 3 follicular lymphoma (FL)
* Ineligible for or have previously received an autologous stem cell transplant (ASCT)
* Relapsed following receipt of the last dose of systemic chemotherapy or ASCT
* At least one prior chemotherapy regimen. Prior chemotherapy regimen must have contained anthracycline (unless contraindicated)
* If the subject is female, she must be non-pregnant and non-lactating at the Baseline Visit. All sexually active males and females of childbearing potential must agree to use an adequate method of contraception throughout the study period
* Eastern Cooperative Oncology Group (ECOG) performance status </= 1

Exclusion Criteria:

* Use of any standard/experimental anti-lymphoma drug therapy within 21 days of the Baseline Visit
* Use of systemic steroids within 5 days of the Baseline Visit (except for the purposes of pre-medication prior to study regimen treatment)
* Prior allogeneic stem cell transplant (SCT)
* The subject has been previously treated with YM155
* The subject has known human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C antibody
* The subject has received other investigational therapy or procedures within 21 days prior to the first study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate (Confirmed Complete Remission +Confirmed Partial Remission) | After the last non-progressing subject receives 8 cycles of treatment or discontinues the treatment

SECONDARY OUTCOMES:
Confirmed Complete remission rate | After the last non-progressing subject receives 8 cycles of treatment or discontinues the treatment
Confirmed Partial remission rate | After the last non-progressing subject receives 8 cycles of treatment or discontinues the treatment
Time to response | After the last non-progressing subject receives 8 cycles of treatment or discontinues the treatment
Duration of response | After the last non-progressing subject receives 8 cycles of treatment or discontinues the treatment
Clinical benefit rate | After the last non-progressing subject receives 8 cycles of treatment or discontinues the treatment
Progression-free survival | After the last non-progressing subject receives 8 cycles of treatment or discontinues the treatment
Overall survival | 1 year after the last subject completes treatment
Safety assessed by recording of adverse events, physical examinations, vital signs, laboratory assessments and electrocardiograms (ECGs) | After the last non-progressing subject receives 8 cycles of treatment or discontinues the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (19):
- United States (6):
  - Site US2778 John B. Amos Cancer Center, Columbus, Georgia
  - Site US55 Loyola University Hospital - Maywood, Maywood, Illinois
  - Site US9 Mount Sinai School of Medicine, New York, New York
  - Site US2802 Mecklenburg Medical Group, Charlotte, North Carolina
  - Site US2149 Gabrail Cancer Center Research, Canton, Ohio
  - Site US402 University of Texas Health Science Center - San Antonio, San Antonio, Texas
- France (5):
  - Site FR1926 Institut Bergonie, Bordeaux
  - Site FR2700 Centre Antoine Lacassagne, Nice
  - Site FR476 Hopital Saint Louis, Paris
  - Site FR1889 Centre de Lutte Contre le Cancer - Centre Henri Becquerel, Rouen
  - Site FR1897 Hopital Bretonneau, Tours
- Spain (4):
  - Site ES1349 Hospital del Mar, Barcelona
  - Site ES1339 Hospital Universitario Ramon y Cajal, Madrid
  - Site ES2967 Hosptial Universitario Madrid Sanchinarro, Madrid
  - Site ES1346 Hospital Universitario de Salamanca, Salamanca
- United Kingdom (4):
  - Site GB2702 Addenbrookes Hospital, Cambridge
  - Site GB1928 St. Georges Hospital, London
  - Site GB2624 The Christie NHS Foundation Trust, Manchester
  - Site GB1903 Oxford Radcliffe Hospital, Oxford